CLINICAL TRIAL: NCT03967223
Title: Master Protocol to Assess the Safety and Antitumor Activity of Genetically Engineered NY-ESO-1-Specific (c259) T Cells, Alone or in Combination With Other Agents, in HLA-A2+ Participants With NY-ESO-1 and/or LAGE-1a Positive Solid Tumors (IGNYTE-ESO)
Brief Title: Master Protocol to Assess the Safety and Antitumor Activity of Genetically Engineered T Cells in NY-ESO-1 and/or LAGE-1a Positive Solid Tumors
Acronym: IGNYTE-ESO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 208467
Record Dates: First submitted 2019-05-10; First posted 2019-05-30 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-10

CONDITIONS: Neoplasms
Keywords: Adoptive T-cell therapy; Advanced metastatic disease; Advanced unresectable disease; Synovial sarcoma; Myxoid/round cell liposarcoma; GSK3377794; Positive solid tumors; T-cell receptors; Leukapheresis; Letetresgene autoleucel; Lete-cel
MeSH Terms: conditions — Neoplasms; Sarcoma, Synovial; Liposarcoma, Myxoid | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Masking Description: This will be an open-label study. Hence, there will be no masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Substudy 1: lete-cel in previously untreated advanced (metastatic or unresectable) SS or MRCLS (Experimental): Eligible participants will be leukapheresed to manufacture engineered T cells. Participants will then receive letetresgene autoleucel.
  Interventions: Drug: Letetresgene autoleucel (lete-cel, GSK3377794); Drug: Fludarabine; Drug: Cyclophosphamide
- Substudy 2: lete-cel in advanced (metastatic or unresectable) SS or MRCLS post anthracycline chemo (Experimental): Eligible participants will be leukapheresed to manufacture engineered T cells. Participants will then receive letetresgene autoleucel.
  Interventions: Drug: Letetresgene autoleucel (lete-cel, GSK3377794); Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Letetresgene autoleucel (lete-cel, GSK3377794) — letetresgene autoleucel will be administered.
Drug: Fludarabine — Fludarabine will be used as the lymphodepleting chemotherapy
Drug: Cyclophosphamide — Cyclophosphamide will be used as the lymphodepleting chemotherapy.

SUMMARY:
This trial will evaluate safety and efficacy of human engineered T-cell therapies, in participants with advanced tumors.

DETAILED DESCRIPTION:
New York esophageal antigen-1 (NY-ESO-1) and LAGE-1a antigens are tumor-associated proteins that have been found in several tumor types. Clinical trials using adoptively transferred T cells directed against NY-ESO-1/LAGE-1a have shown objective responses. Letetresgene autoleucel (lete-cel, GSK3377794) is the first generation of NY-ESO-1 specific T-cell receptor engineered T cells. This is a master protocol investigating T-cell therapies. It will initially consist of a core protocol with two independent substudies investigating Letetresgene autoleucel in previously untreated (1L) Human Leukocyte Antigen (HLA)-A*02+ participants with NY-ESO-1+ advanced (metastatic or unresectable) synovial sarcoma (SS) or myxoid/round cell liposarcoma (MRCLS) (Substudy 1) and Letetresgene autoleucel as second line or higher (2L+) treatment in HLA-A*02+ participants with NY-ESO-1+ advanced (metastatic or unresectable) SS or MRCLS who have progressed following treatment with anthracycline based chemotherapy (Substudy 2).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be greater than or equal to 10 years of age on the day of signing informed consent.
* Participant scheduled to receive clinical drug product supply must also weigh ≥40 kg
* Participant must be positive for HLA-A*02:01, HLA-A*02:05, and/or HLA-A*02:06 alleles by a designated central laboratory
* Participant's tumor is positive for NY-ESO-1 expression by a designated central laboratory.
* Participant has a diagnosis of synovial sarcoma (SS) or myxoid/round cell liposarcoma (MRCLS)
* Performance status: dependent on age - Lansky > 60, Karnofsky > 60, Eastern Cooperative Oncology Group 0-1.
* Participant must have adequate organ function and blood cell counts, within 7 days prior to leukapheresis.
* At time of treatment, participant has measurable disease according to RECIST v1.1.
* Male or female. Contraception requirements will apply at the time of leukapheresis and treatment.
* Consultation for prior history per protocol specifications.

Exclusion Criteria:

* Central nervous system metastases.
* Any other prior malignancy that is not in complete remission.
* Clinically significant systemic illness (Serious active infections or significant cardiac, pulmonary, hepatic or other organ dysfunction, that in the judgment of the Investigator would compromise the participant's ability to tolerate protocol therapy or significantly increase the risk of complications).
* Prior or active demyelinating disease.
* History of chronic or recurrent (within the last year prior to leukapheresis) severe autoimmune or immune mediated disease (e.g. Crohn's disease, systemic lupus) requiring steroids or other immunosuppressive treatments.
* Previous treatment with genetically engineered NY-ESO-1-specific T cells.
* Previous NY-ESO-1 vaccine or NY-ESO-1 targeting antibody.
* Prior gene therapy using an integrating vector.
* Previous allogeneic hematopoietic stem cell transplant.
* Washout periods for prior radiotherapy and systemic chemotherapy must be followed.
* Participant had major surgery in less than or equal to 28 days of first dose of study intervention.
* Prior radiation exceeds protocol specified limits.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Substudy 1: Overall response rate (ORR) | Until disease progression (up to 5 years)
  Overall response rate is defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) relative to the total number of participants within the analysis population at any time per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. as determined by the local investigators.
Substudy 2: Overall response rate (ORR) as assessed by central independent review | Up to 5 years
  Overall response rate is defined as the percentage of participants with a confirmed CR or PR relative to the total number of participants within the analysis population at any time per RECIST v1.1. as assessed by central independent review.

SECONDARY OUTCOMES:
Substudy 1 and 2: Time to response (TTR) | Until disease progression (up to 5 years)
  Time to response is defined as time from date of T-cell administration to first documented evidence of confirmed (CR or PR) as assessed by local investigators per RECIST v1.1.
Substudy 1 and 2: Duration of response (DOR) | Until disease progression (up to 5 years)
  Duration of response is defined as, in the subset of participants who show a confirmed CR or PR as assessed by local investigators, the time from first documented evidence of CR or PR until the first documented sign of disease progression or death.
Substudy 1 and 2: Disease control rate (DCR) | Until disease progression (up to 5 years)
  Disease control rate is defined as the percentage of participants with a confirmed CR, PR, or stable disease (SD) with minimal 12 weeks duration relative to the total number of participants within the analysis population at the time of primary analysis as determined by Investigators per RECIST v1.1.
Substudy 1 and 2: Progression free survival (PFS) | Until disease progression (up to 5 years)
  Progression free survival is defined as the time from the date of T-cell administration until first documented sign of disease progression per RECIST v1.1, or death.
Substudy 1 and 2: Frequency of adverse events (AEs), serious adverse events (SAEs) and AEs of special interest (AESI) according to severity | Until disease progression (up to 5 years)
  AEs, SAEs and AESIs will be collected. Severity of AEs and SAEs will be summarized using National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.
Substudy 1 and 2: Number of participants with replication competent lentivirus (RCL) | Until disease progression (up to 5 years)
  RCL exposure will be assessed by polymerase chain reaction (PCR) based assay.
Substudy 1 and 2: Number of participants with insertional oncogenesis (IO) | Until disease progression (up to 5 years)
  Peripheral blood mononuclear cells (PBMC) samples will be collected for monitoring insertional oncogenesis by PCR for gene modified cells in the blood.
Substudy 2: Number of participants with clinically significant changes in hematology, clinical chemistry and urinalysis parameters | Until disease progression (up to 5 years)
  Blood and urine samples will be collected for assessment of hematology, clinical chemistry and urinalysis parameters.
Substudy 1 and 2: Maximum transgene expansion (Cmax) of letetresgene autoleucel | Until disease progression (up to 5 years)
  Whole blood samples will be collected at indicated time points for evaluation of Cmax.
Substudy 1 and 2: Time to Cmax (Tmax) of letetresgene autoleucel | Until disease progression (up to 5 years)
  Whole blood samples will be collected at indicated time points for evaluation of Tmax.
Substudy 1 and 2: Area under the concentration/persistence time curve from zero to time t (AUC[0-t]) of letetresgene autoleucel | Until disease progression (up to 5 years)
  Whole blood samples will be collected at indicated time points for evaluation of AUC(0-t).
Substudy 2: Overall response rate (ORR) as determined by the local investigators | Up to 5 years
  Overall response rate is defined as the percentage of participants with a confirmed CR or PR relative to the total number of participants within the analysis population at any time per RECIST v1.1. as determined by the local investigators.
Substudy 2: Overall Survival (OS) | Up to 5 years
  Overall Survival is defined as the interval of time between the date of T-cell infusion and the date of death.
Substudy 2: Number of participants with positive anti-drug antibodies (ADA) and titers of ADA against letetresgene autoleucel | Up to 36 months
  Serum samples will be collected to analyze for the presence of ADAs using validated immunoassays.

CONTACTS AND LOCATIONS:
Overall Officials: Adaptimmune, Study Director — Adaptimmune
Locations (38):
- United States (24):
  - City of Hope National Medical Center, Duarte, California
  - Stanford Hospital and Clinics, Stanford, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - University of Iowa College of Medicine, Iowa City, Iowa
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering cancer center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University-Columbus, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh, Hillman Cancer Centre, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University Of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research, Seattle, Washington
  - Froedtert Hospital, Milwaukee, Wisconsin
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CIUSSS de L'Est-De-Lile-De-Montreal, Montreal, Quebec
- France (2):
  - Centre Léon Bérard, Lyon
  - CHU de Bordeaux GH Sud Hôpital Haut Lévêque, Pessac
- Italy (2):
  - Fondazione IRCCS Instituto Nazionale Dei Tumori, Milan, Lombardy
  - Ircss Istituto Clinico Humanitas, Rozzano (MI), Lombardy
- The Netherlands Cancer Institute, Amsterdam, Netherlands
- Spain (4):
  - Hospital Santa Creu Y Sant Pau, Barcelona
  - Ico Duran y Reynals l'Hospitalet de Llobrega, Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Virgen Del Rocio, Seville
- United Kingdom (3):
  - Royal Marsden Hospital, London
  - University College Hospital-London, London
  - Christie Hospital NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No